CLINICAL TRIAL: NCT04255485
Title: Long Term Neurobehavioral Effects of Anesthetics and Cochlear Implantation on Infants With Hearing Impairment
Brief Title: The Neurobehavioral Effects of Anesthetics on Infants With Hearing Impairment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Jingjie Li, associate chief physician, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: SH9H-2019-T19-2
Record Dates: First submitted 2020-01-26; First posted 2020-02-05 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Long Term Neurobehavioral Effects
Keywords: infant; anesthesia; neurobehavioral development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Short time anesthesia group: Unilateral cochlear implantation,which time of anesthesia is less than 3 hours
- Long time anesthesia group: Bilateral cochlear implantation, which time of anesthesia is more than 3 hours

SUMMARY:
The long-term effect of general anesthesia on developing brain is the focus of clinicians when infants exposed to general anesthesia for a long time during operation. A retrospective study showed that children exposed to long-term or repeated operations, the anesthetics had a higher incidence of cognitive impairment in adolescence than those did no. When infants with hearing impairment undergo bilateral cochlear implant surgery, they are at high risk of long-term neurobehavioral abnormalities caused by anesthesia. In this study, investigators intend to observe the long-term behavioral abnormalities of hearing-impaired infants after unilateral or bilateral cochlear implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Infants aged between 6 months and 2 years old undergoing cochlear implantation under general anesthesia in 9th hospital
2. Patients who have not participated in other clinical trials
3. ASA class I-II selective operation without any acute infectious diseases or systematic diseases
4. Infant's family members agree to participated in the trials and sign the informed consent

Exclusion Criteria:

1. Reject to sign the informed consent and participate in the trials
2. Patients with severe liver and kidney damage or other heart, lung and nervous system diseases
3. The Gesell developmental scale is less than 86 in motor behavior and physical energy
4. With a history of intrauterine distress, umbilical cord around the neck, hypoxia and jaundice
5. Infant who is allergic to egg and milk
6. Family history of malignant hyperthermia
7. Allergy to anesthetic drugs

Ages: 6 Months to 2 Years | Sex: All
Age Groups: Child
Study Population: Children undergoing cochlear implantation under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2019-04-08 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
change of Baseline Gesell Developmental Scale after 6 month | change in 6 months after surgery
  Neurobehavior effects

SECONDARY OUTCOMES:
change of Baseline Gesell Developmental Scale after 12 month | change in 12 months after surgery
  Neurobehavior effects

CONTACTS AND LOCATIONS:
Overall Officials: Jingjie Li, M.D, Study Chair — Shanghai No.9 People's Hospital
Locations (1):
- Shanghai No.9 People's Hospital, Shanghai, China

DOCUMENTS (1):
  • Informed Consent Form (2019-01-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT04255485/ICF_001.pdf